CLINICAL TRIAL: NCT05572931
Title: Effect of Fu's Subcutaneous Needling on Postoperative Acute Pain in Patients With Lumbar Spine Surgery: a Single-blinded Randomized, Control Study
Brief Title: Effect of Fu's Subcutaneous Needling on Postoperative Acute Pain in Patients With Lumbar Spine Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Ying Wu, Attending physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH109-REC2-116
Record Dates: First submitted 2022-10-02; First posted 2022-10-10 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative
Keywords: Fu's Subcutaneous Needling, postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham comparator (Sham Comparator): In addition to the routine analgesic (Acetaminophen 500mg, TID), the patients were treated with sham FSN at the 1st, 24th, and 48th hours after surgery. The sham FSN was used a fine acupuncture needle without swaying movement and reperfusion approach.
  Interventions: Device: fine acupuncture needle
- Experimental (Experimental): In addition to postoperative routine analgesic (Acetaminophen 500mg, TID), patients were received FSN treatment. The FSN insertion point and time are the same as control group. And then we performed swaying movement and reperfusion approach.
  Interventions: Device: Fu's Subcutaneous Needling(FSN)

INTERVENTIONS:
Device: Fu's Subcutaneous Needling(FSN) — Insertion points are both sides of 1) inferior edge of the scapula; 2)the midpoint of inferior edge of the posterior superior iliac spine and the ischial tuberosity.
  FSN (Trocar Acupuncture Needle, Nanjing FSN Medical Co. , Ltd, China.) ) is a solid needle with plastic cannula tube on the outside. Add on swaying movement (SM) and reperfusion approach (RA) after the needle inserting into the subcutaneous layer. The SM is a horizontal fan sway movement with the base of the needle for the fulcrum, The SM speed is 200 times in 2 minutes. Apply RA when performing SM. RA movement is hip extension in prone position with resistance by physician's hand for 10 seconds. And then rest for 10 seconds. Repeat 3 cycles. The same RA is performed over the other three insertion point.
  Arms: Experimental
Device: fine acupuncture needle — (36G, 0.5 inch, Wujiang city cloud & dragon medical device Co.,Ltd.) Only inserted to skin, not into the subcutaneous layer. No SM and RA.
  Arms: Sham comparator

SUMMARY:
The goal of this clinical trial is to evaluate Fu's Subcutaneous Needling (FSN) in postoperative pain in patients with Lumbar Spine Surgery (LSS). The main questions it aims to answer are:

* Is FSN effective for postoperative pain?
* Dose FSN decrease the tissue hardness after LSS?
* Dose FSN have the effect of anti-inflammatory after LSS?

Participants will receive routine analgesic and FSN after LSS. Researchers will compare Sham group to see if FSN being effective for postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Pain and neurological symptoms are caused by degeneration of the spine (L1-S1) and require surgery.
* One hour after lumbar spine surgery (evaluated after returning to the ward from the recovery room) Visual analogue scale (VAS) score ≥ 5 points
* After being explained, join the trial voluntarily and sign the subject's consent form.

Exclusion Criteria:

* Pain caused by acute trauma.
* major diseases such as heart and lung failure, cancer, chronic kidney disease.
* psychiatric disorder.
* History of substance abuse.
* A history of spinal surgery.
* Refused sign the consent form.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Change of Taiwanese version of the Brief Pain Inventory (BPI-T) Short Form | Change from Baseline BPI-T at the 1st、24th、48th、72nd hour after surgery.
  BPI-T Short Form
The total dosage of analgesic drug | The amount of intravenous opioid drug (Pethidine 50mg/vail) within 72 hours after surgery.
  opioid drug (Pethidine 50mg/vail)

SECONDARY OUTCOMES:
Change of Blood serum C-reactive protein (CRP) | Change from Baseline CRP at the 24th, 72nd hour, 1st month after surgery.
  Biochemistry
Change of Blood serum IL-1ẞ、IL-2、IL-6 | Change from Baseline IL-1ẞ、IL-2、IL-6 at the 24th, 72nd hour, 1st month after surgery.
  Biochemistry
Change of Blood serum TNF-α | Change from Baseline TNF-α at the 24th, 72nd hour, 1st month after surgery.
  Biochemistry
Change of Tissue hardness (TH) | Change from Baseline TH at the 1st、24th、48th、72nd hour after surgery.
  The points for measuring TH were the inferior border of the scapula, two centimeters horizontal from the midline of the L3 level, and the gluteus maximus.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ying Wu, MD, Study Chair — China Medical University, China
Locations (1):
- China Medical University Hsinchu Hospital, Zhubei, Hsinchu County, Taiwan

IPD SHARING:
Plan to Share IPD: No